CLINICAL TRIAL: NCT06781229
Title: Non-interventional Study Exploring the Composition of the Periodontal Microbiota of Patients with Body Mass Index Greater Than 30 That Are Candidates for Bariatric Surgery
Brief Title: Periodontal Microbiota of Patients Candidates for Bariatric Surgery with Body Mass Index Greater Than 30
Acronym: OROBESITE
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/24/0432
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Bariatric Surgery; Obesity, Morbid
Keywords: microbiological composition; obese; bypass; Body mass index
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * 5g of visceral adipose tissue and 5g of subcutaneous adipose tissue
  * Saliva samples
  * Samples of periodontal plaque in the periodontal sulcus (assessed during partial probing) using sterile paper points (minimum 3 and maximum 10 per patient) inserted for 30 seconds into the periodontal sulcus.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1 : obesity : 30 ≤ BMI < 35: Obese patients with 30 ≤ BMI < 35
- Group 2 : morbid obesity : 35 ≤ BMI: Morbid obese patients with 35 ≤ BMI

SUMMARY:
The goal of this observational study is to compare the microbiological composition of the periodontal plaque of obese people undergoing bariatric surgery according to their Body Mass Index. The main question it aims to answer is:

Does obese patients have different microbiote according to their obesity?

Obesity being classified in two groups :

* group "obesity" for a BMI between 30 and 35
* versus "morbid obesity" group with a BMIabove 35.

Participants who are scheduled to undergo bariatric surgery as part of their regular medical care will answer questions about their quality of life, hygiene habits, and saliva and periodontal samples will be taken.

DETAILED DESCRIPTION:
The study is a non-interventional, single-centre, cross-sectional, comparative study with prospective and consecutive recruitment of participants.

Participants who are scheduled to undergo bariatric surgery as part of their regular medical care will

1. during the odontological visit of approximately one hour:

   * complete standard odontology medical questionnaire
   * complete the dietary hygiene questionnaire: "Etude Nationale Nutrition Santé" questionnaire
   * complete 2 quality of life questionnaires: EQ-5D-5L questionnaire and GOHAI self-questionnaire
   * undergo clinical examination (visual examination and partial periodontal probing),
   * Radiological check-up (panoramic X-ray) and biological check-up (salivary and periodontal samples (non-invasive).
2. During bariatric surgery, surgical techniques create surgical waste. From this operative waste, fragments of visceral adipose tissue may be recovered and, if the surgery so requires, subcutaneous adipose tissue (quantity recovered: 5g of visceral adipose tissue and 5g of subcutaneous adipose tissue). The samples taken will be stored in a hospital tissue bank with a view to possible future re-use. Each patient will be informed of this during the inclusion visit.

ELIGIBILITY:
Inclusion Criteria:

* BMI greater than or equal to 30
* Be on the list of patients scheduled for bariatric surgery,
* Be able to receive information about the study and understand the information form in order to take part in the study. This implies mastering the French language,

Exclusion Criteria:

* Alcohol consumption >30g/d (men) or 20g/d (women),
* Having taken antibiotics, prebiotics or probiotics in the month prior to inclusion (this has an influence on the composition of the patient's microbiota),
* During pregnancy or breastfeeding,
* For whom oral surgery is planned (surgery for benign or malignant tumours of the maxillary and mandibular bone bases), or with a history of oral surgery in the month prior to inclusion,
* At risk of infection (existence of one or more of the following known chronic infectious diseases: HIV, HBV, HCV and mononucleosis) and/or chronic renal insufficiency (creatinine clearance < 60ml/min),
* Patients with a general pathology that contraindicates the performance of diagnostic procedures such as periodontal probing (patients at high risk of infective endocarditis according to the ANSM).
* Totally edentulous patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients scheduled to undergo bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2029-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Taxonomic analysis | before bariatric surgery
  Taxonomic analysis of the microbiological composition of the periodontal plaque between group 1 (obesity) and 2 (morbid obesity) : relative quantities of periodontal bacteria between group 1 (obesity) and 2 (morbid obesity)